CLINICAL TRIAL: NCT06469086
Title: Clinical Significance of Appendicoliths in Conservative Treatment of Acute Complicated Appendicitis Patients With Abscess: A Single-center Retrospective Study
Brief Title: Appendicoliths in Acute Complicated Appendicitis Patients With Abscess
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhongshan-HHY-05
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Acute Complicated Appendicitis With Abscess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical data collection — The clinical significance of appendicoliths in the conservative management of acute complicated appendicitis with abscesses.

SUMMARY:
Complicated appendicitis, characterized by the presence of an abscess or perforation, involves acute inflammation of the peritoneum secondary to an infection of the appendix, presenting additional challenges for management. Traditionally, the standard treatment for complicated appendicitis has been surgical intervention. However, conservative management, involving antibiotics and drainage, has emerged as a viable alternative for selected patients. Recent studies emphasize the importance of selecting appropriate antibiotics based on local resistance patterns and the patient's clinical condition. Broad-spectrum antibiotics, including those targeting anaerobic bacteria, are often preferred. In addition, advances in imaging technology, such as ultrasound-guided drainage, have improved the precision and success rates of percutaneous abscess drainage. This minimally invasive approach helps manage localized infections and can prevent the need for immediate surgery.

One factor that has gained significant attention in determining the success of conservative treatment for acute complicated appendicitis is the presence of appendicoliths-calcified deposits within the appendix. This study aims to investigate the clinical significance of appendicoliths in the conservative management of acute complicated appendicitis with abscesses.

ELIGIBILITY:
Inclusion Criteria:

* Patients who aged ≥18 years, who diagnosed as acute appendicitis clinically, who had peri-appendiceal abscess larger than 2 cm in diameter on CT scan, who agreed conservative treatment first, who refused immediate emergency surgery

Exclusion Criteria:

* Patients younger than 18 years, those with malignancies, those with incomplete clinical or pathological records were excluded from the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute complicated appendicitis patients with absces swho met the criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of conservative treatment | January 01, 2025 to December 31, 2025.

SECONDARY OUTCOMES:
Postoperative complications | January 01, 2025 to December 31, 2025.
Length of postoperative hospital stay | January 01, 2025 to December 31, 2025.
The surgical approach used | January 01, 2025 to December 31, 2025.